CLINICAL TRIAL: NCT02063828
Title: Reducing Lung Cancer-Related Anxiety (RELAX)
Acronym: RELAX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Took too long to accrue participants, stopped for feasibility concerns
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB00038743; U10CA081851 (NIH); WF-01213 (Other: NCI); 1UG1CA189824 (NIH); 2R25CA122061-07 (NIH); R21CA182111-01 (NIH); NCI-2014-02413 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-01-27; First posted 2014-02-14 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer
Keywords: anxiety; Dyspnea; respiratory functioning
MeSH Terms: conditions — Lung Neoplasms; Anxiety Disorders; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group A (Experimental): Group A - Device Guided Breathing Low Dose
  Interventions: Device: Group A - Device guided breathing low dose
- Group B (Experimental): Group B - Device guided breathing high dose
  Interventions: Device: Group B - Device guided breathing high dose
- Group C (Sham Comparator): Group C - Usual Breathing Control Group
  Interventions: Device: Group C - Usual Breathing Control Group

INTERVENTIONS:
Device: Group A - Device guided breathing low dose — Group A: 15 minutes once a day, 5 days a week for 12 weeks.
  Other Names: RESPeRATE (InterCure Ltd) Device
  Arms: Group A
Device: Group B - Device guided breathing high dose — Group B - 15 minutes twice a day, 5 days a week for 12 weeks.
  Other Names: RESPeRATE (InterCure Ltd) Device
  Arms: Group B
Device: Group C - Usual Breathing Control Group — Group C - 15 minutes per day, 5 days a week for 12 weeks.
  Other Names: RESPeRATE (InterCure Ltd) Device
  Arms: Group C

SUMMARY:
The purpose of this research study is to compare the effects of music and different levels of device-guided breathing on anxiety and shortness of breath in lung cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES

1. To assess feasibility (accrual, participation, adherence, retention) of a randomized study of device-guided breathing and music in 75 post-treatment lung cancer survivors with significant anxiety.
2. To obtain preliminary data on the variability and efficacy of two doses of a device-guided breathing intervention versus a music control group for reducing anxiety (primary outcome) and for improving self-reported dyspnea and respiratory functioning (secondary outcomes) in post-treatment lung cancer survivors.
3. To select the optimal dose of the device-guided breathing intervention (15 minutes once/day or twice/day) for subsequent randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Past History of any lung cancer
* For Stage I-III disease, patients should be 2-24 months post-completion of surgery, radiation therapy and/or chemotherapy with no further planned treatment during the 12-week study and no evidence of disease.
* For Stage IV disease, patients may be receiving no treatment or may be receiving maintenance treatment with a target agent, chemotherapy, or immunotherapy provided the most recent imaging does not demonstrate progressive disease.
* After completion of all three screening questionnaires, participant must score accordingly on at least one questionnaire to be eligible.
* Willing/able to attend brief introductory session and use assigned device for the assigned period of time (15 minutes once or twice per day), at least 5 days per week for 12 weeks
* Age ≥ 18 years
* Must have telephone

Exclusion Criteria:

* Patient does not understand English
* Active lung infection
* Progressive cancer (must be considered no evidence of disease or stable)
* Any change in psychotropic medications in past 30 days
* Hearing loss that would preclude participating in interventions. Adequate hearing to participate will be determined via: (1) Response of "no" to the question ["Do you have a hearing problem now?"] Participants with hearing aids will be allowed to enroll as long as their hearing is adequate to hear the sounds on the study devices. If necessary, potential study participants will receive a brief test trial with the RESPeRATE device. If they indicate inability to hear the guiding tones, they will not be enrolled in the study.

Cortisol Exclusion

- Participants with endocrine disorders (e.g., diabetes and thyroid disorders) or on steroid-based medications are excluded from the cortisol portion of the study (with the exception of topical hydrocortisone that is permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C Danhauer, PhD, Study Chair — Wake Forest University Health Sciences; Glenn Lesser, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (11):
- United States (11):
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pal GK, Velkumary S, Madanmohan. Effect of short-term practice of breathing exercises on autonomic functions in normal human volunteers. Indian J Med Res. 2004 Aug;120(2):115-21. PMID 15347862
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Bach PB, Mirkin JN, Oliver TK, Azzoli CG, Berry DA, Brawley OW, Byers T, Colditz GA, Gould MK, Jett JR, Sabichi AL, Smith-Bindman R, Wood DE, Qaseem A, Detterbeck FC. Benefits and harms of CT screening for lung cancer: a systematic review. JAMA. 2012 Jun 13;307(22):2418-29. doi: 10.1001/jama.2012.5521. PMID 22610500
- [Background] Wender R, Fontham ET, Barrera E Jr, Colditz GA, Church TR, Ettinger DS, Etzioni R, Flowers CR, Gazelle GS, Kelsey DK, LaMonte SJ, Michaelson JS, Oeffinger KC, Shih YC, Sullivan DC, Travis W, Walter L, Wolf AM, Brawley OW, Smith RA. American Cancer Society lung cancer screening guidelines. CA Cancer J Clin. 2013 Mar-Apr;63(2):107-17. doi: 10.3322/caac.21172. Epub 2013 Jan 11. PMID 23315954
- [Background] Doria-Rose VP, White MC, Klabunde CN, Nadel MR, Richards TB, McNeel TS, Rodriguez JL, Marcus PM. Use of lung cancer screening tests in the United States: results from the 2010 National Health Interview Survey. Cancer Epidemiol Biomarkers Prev. 2012 Jul;21(7):1049-59. doi: 10.1158/1055-9965.EPI-12-0343. Epub 2012 May 9. PMID 22573798
- [Background] Alfano CM, Rowland JH. Recovery issues in cancer survivorship: a new challenge for supportive care. Cancer J. 2006 Sep-Oct;12(5):432-43. doi: 10.1097/00130404-200609000-00012. PMID 17034679
- [Background] Hodgkinson K, Butow P, Fuchs A, Hunt GE, Stenlake A, Hobbs KM, Brand A, Wain G. Long-term survival from gynecologic cancer: psychosocial outcomes, supportive care needs and positive outcomes. Gynecol Oncol. 2007 Feb;104(2):381-9. doi: 10.1016/j.ygyno.2006.08.036. Epub 2006 Oct 5. PMID 17027072
- [Background] Jacobsen PB DKSZetal. Management of anxiety and depression in adult cancer patients: Toward an evidence-based approach. In: Chang AE GPHDea, editor. Oncology: An Evidence-Based Approach. Philadelphia, PA: Springer; 2006. p. 1552-79.
- [Background] Jefford M, Karahalios E, Pollard A, Baravelli C, Carey M, Franklin J, Aranda S, Schofield P. Survivorship issues following treatment completion--results from focus groups with Australian cancer survivors and health professionals. J Cancer Surviv. 2008 Mar;2(1):20-32. doi: 10.1007/s11764-008-0043-4. Epub 2008 Jan 25. PMID 18648984
- [Background] Stanton AL, Bower JE, Low CA. Posttraumatic Growth After Cancer. In 2006. p. 138-75.
- [Background] Brintzenhofe-Szoc KM, Levin TT, Li Y, Kissane DW, Zabora JR. Mixed anxiety/depression symptoms in a large cancer cohort: prevalence by cancer type. Psychosomatics. 2009 Jul-Aug;50(4):383-91. doi: 10.1176/appi.psy.50.4.383. PMID 19687179
- [Background] Zabora J, BrintzenhofeSzoc K, Curbow B, Hooker C, Piantadosi S. The prevalence of psychological distress by cancer site. Psychooncology. 2001 Jan-Feb;10(1):19-28. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-6. PMID 11180574
- [Background] Li J, Girgis A. Supportive care needs: are patients with lung cancer a neglected population? Psychooncology. 2006 Jun;15(6):509-16. doi: 10.1002/pon.983. PMID 16292789
- [Background] Baker F, Denniston M, Smith T, West MM. Adult cancer survivors: how are they faring? Cancer. 2005 Dec 1;104(11 Suppl):2565-76. doi: 10.1002/cncr.21488. PMID 16258929
- [Background] Uchitomi Y, Mikami I, Nagai K, Nishiwaki Y, Akechi T, Okamura H. Depression and psychological distress in patients during the year after curative resection of non-small-cell lung cancer. J Clin Oncol. 2003 Jan 1;21(1):69-77. doi: 10.1200/JCO.2003.12.139. PMID 12506173
- [Background] Ostroff JS, Krebs P, Coups EJ, Burkhalter JE, Feinstein MB, Steingart RM, Logue AE, Park BJ. Health-related quality of life among early-stage, non-small cell, lung cancer survivors. Lung Cancer. 2011 Jan;71(1):103-8. doi: 10.1016/j.lungcan.2010.04.011. Epub 2010 May 11. PMID 20462654
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Hung R, Krebs P, Coups EJ, Feinstein MB, Park BJ, Burkhalter J, Ostroff JS. Fatigue and functional impairment in early-stage non-small cell lung cancer survivors. J Pain Symptom Manage. 2011 Feb;41(2):426-35. doi: 10.1016/j.jpainsymman.2010.05.017. Epub 2011 Jan 8. PMID 21216563
- [Background] Linden W, Vodermaier A, Mackenzie R, Greig D. Anxiety and depression after cancer diagnosis: prevalence rates by cancer type, gender, and age. J Affect Disord. 2012 Dec 10;141(2-3):343-51. doi: 10.1016/j.jad.2012.03.025. Epub 2012 Jun 21. PMID 22727334
- [Background] Smith EL, Hann DM, Ahles TA, Furstenberg CT, Mitchell TA, Meyer L, Maurer LH, Rigas J, Hammond S. Dyspnea, anxiety, body consciousness, and quality of life in patients with lung cancer. J Pain Symptom Manage. 2001 Apr;21(4):323-9. doi: 10.1016/s0885-3924(01)00255-x. PMID 11312047
- [Background] Tanaka K, Akechi T, Okuyama T, Nishiwaki Y, Uchitomi Y. Prevalence and screening of dyspnea interfering with daily life activities in ambulatory patients with advanced lung cancer. J Pain Symptom Manage. 2002 Jun;23(6):484-9. doi: 10.1016/s0885-3924(02)00394-9. PMID 12067772
- [Background] Dudgeon DJ, Lertzman M, Askew GR. Physiological changes and clinical correlations of dyspnea in cancer outpatients. J Pain Symptom Manage. 2001 May;21(5):373-9. doi: 10.1016/s0885-3924(01)00278-0. PMID 11369157
- [Background] Henoch I, Bergman B, Danielson E. Dyspnea experience and management strategies in patients with lung cancer. Psychooncology. 2008 Jul;17(7):709-15. doi: 10.1002/pon.1304. PMID 18074408
- [Background] Ryan LS. Psychosocial issues and lung cancer: a behavioral approach. Semin Oncol Nurs. 1996 Nov;12(4):318-23. doi: 10.1016/s0749-2081(96)80031-3. PMID 8936648
- [Background] Hopwood P, Stephens RJ. Symptoms at presentation for treatment in patients with lung cancer: implications for the evaluation of palliative treatment. The Medical Research Council (MRC) Lung Cancer Working Party. Br J Cancer. 1995 Mar;71(3):633-6. doi: 10.1038/bjc.1995.124. PMID 7533520
- [Background] Muers MF, Round CE. Palliation of symptoms in non-small cell lung cancer: a study by the Yorkshire Regional Cancer Organisation Thoracic Group. Thorax. 1993 Apr;48(4):339-43. doi: 10.1136/thx.48.4.339. PMID 7685550
- [Background] Reuben DB, Mor V. Dyspnea in terminally ill cancer patients. Chest. 1986 Feb;89(2):234-6. doi: 10.1378/chest.89.2.234. PMID 3943383
- [Background] Sarna L, Evangelista L, Tashkin D, Padilla G, Holmes C, Brecht ML, Grannis F. Impact of respiratory symptoms and pulmonary function on quality of life of long-term survivors of non-small cell lung cancer. Chest. 2004 Feb;125(2):439-45. doi: 10.1378/chest.125.2.439. PMID 14769722
- [Background] Feinstein MB, Krebs P, Coups EJ, Park BJ, Steingart RM, Burkhalter J, Logue A, Ostroff JS. Current dyspnea among long-term survivors of early-stage non-small cell lung cancer. J Thorac Oncol. 2010 Aug;5(8):1221-6. doi: 10.1097/JTO.0b013e3181df61c8. PMID 20592631
- [Background] Tishelman C, Degner LF, Rudman A, Bertilsson K, Bond R, Broberger E, Doukkali E, Levealahti H. Symptoms in patients with lung carcinoma: distinguishing distress from intensity. Cancer. 2005 Nov 1;104(9):2013-21. doi: 10.1002/cncr.21398. PMID 16178002
- [Background] Tanaka K, Akechi T, Okuyama T, Nishiwaki Y, Uchitomi Y. Factors correlated with dyspnea in advanced lung cancer patients: organic causes and what else? J Pain Symptom Manage. 2002 Jun;23(6):490-500. doi: 10.1016/s0885-3924(02)00400-1. PMID 12067773
- [Background] O'Driscoll M, Corner J, Bailey C. The experience of breathlessness in lung cancer. Eur J Cancer Care (Engl). 1999 Mar;8(1):37-43. doi: 10.1046/j.1365-2354.1999.00129.x. PMID 10362952
- [Background] Gupta D, Lis CG, Grutsch JF. The relationship between dyspnea and patient satisfaction with quality of life in advanced cancer. Support Care Cancer. 2007 May;15(5):533-8. doi: 10.1007/s00520-006-0178-7. Epub 2006 Nov 21. PMID 17120067
- [Background] Wilhelm FH, Gevirtz R, Roth WT. Respiratory dysregulation in anxiety, functional cardiac, and pain disorders. Assessment, phenomenology, and treatment. Behav Modif. 2001 Sep;25(4):513-45. doi: 10.1177/0145445501254003. PMID 11530714
- [Background] Clark ME, Hirschman R. Effects of paced respiration on anxiety reduction in a clinical population. Biofeedback Self Regul. 1990 Sep;15(3):273-84. doi: 10.1007/BF01011109. PMID 2223892
- [Background] Eisen AR, Rapee RM, Barlow DH. The effects of breathing rate and pCO2 levels on relaxation and anxiety in a non-clinical population. Journal of Anxiety Disorders 1990;4(3):183-90
- [Background] Hazlett-Stevens H, Craske MG. BREATHING RETRAINING AND DIAPHRAGMATIC BREATHING. In General principles and empirically supported techniques of cognitive behavior therapy. 2009.
- [Background] Zhao I, Yates P. Non-pharmacological interventions for breathlessness management in patients with lung cancer: a systematic review. Palliat Med. 2008 Sep;22(6):693-701. doi: 10.1177/0269216308095024. PMID 18715967
- [Background] Bredin M, Corner J, Krishnasamy M, Plant H, Bailey C, A'Hern R. Multicentre randomised controlled trial of nursing intervention for breathlessness in patients with lung cancer. BMJ. 1999 Apr 3;318(7188):901-4. doi: 10.1136/bmj.318.7188.901. PMID 10102851
- [Background] Corner J, Plant H, A'Hern R, Bailey C. Non-pharmacological intervention for breathlessness in lung cancer. Palliat Med. 1996 Oct;10(4):299-305. doi: 10.1177/026921639601000405. PMID 8931065
- [Background] Schein MH, Gavish B, Herz M, Rosner-Kahana D, Naveh P, Knishkowy B, Zlotnikov E, Ben-Zvi N, Melmed RN. Treating hypertension with a device that slows and regularises breathing: a randomised, double-blind controlled study. J Hum Hypertens. 2001 Apr;15(4):271-8. doi: 10.1038/sj.jhh.1001148. PMID 11319676
- [Background] Elliot WJ, Izzo JL Jr, White WB, Rosing DR, Snyder CS, Alter A, Gavish B, Black HR. Graded blood pressure reduction in hypertensive outpatients associated with use of a device to assist with slow breathing. J Clin Hypertens (Greenwich). 2004 Oct;6(10):553-9; quiz 560-1. doi: 10.1111/j.1524-6175.2004.03553.x. PMID 15470284
- [Background] Logtenberg SJ, Kleefstra N, Houweling ST, Groenier KH, Bilo HJ. Effect of device-guided breathing exercises on blood pressure in hypertensive patients with type 2 diabetes mellitus: a randomized controlled trial. J Hypertens. 2007 Jan;25(1):241-6. doi: 10.1097/HJH.0b013e32801040d5. PMID 17143197
- [Background] Meles E, Giannattasio C, Failla M, Gentile G, Capra A, Mancia G. Nonpharmacologic treatment of hypertension by respiratory exercise in the home setting. Am J Hypertens. 2004 Apr;17(4):370-4. doi: 10.1016/j.amjhyper.2003.12.009. PMID 15062893
- [Background] Coups EJ, Ostroff JS. A population-based estimate of the prevalence of behavioral risk factors among adult cancer survivors and noncancer controls. Prev Med. 2005 Jun;40(6):702-11. doi: 10.1016/j.ypmed.2004.09.011. PMID 15850868
- [Background] Grossman E, Grossman A, Schein MH, Zimlichman R, Gavish B. Breathing-control lowers blood pressure. J Hum Hypertens. 2001 Apr;15(4):263-9. doi: 10.1038/sj.jhh.1001147. PMID 11319675
- [Background] Schein MH, Gavish B, Baevsky T, Kaufman M, Levine S, Nessing A, Alter A. Treating hypertension in type II diabetic patients with device-guided breathing: a randomized controlled trial. J Hum Hypertens. 2009 May;23(5):325-31. doi: 10.1038/jhh.2008.135. Epub 2008 Nov 13. PMID 19005477
- [Background] Ekman I, Kjellstrom B, Falk K, Norman J, Swedberg K. Impact of device-guided slow breathing on symptoms of chronic heart failure: a randomized, controlled feasibility study. Eur J Heart Fail. 2011 Sep;13(9):1000-5. doi: 10.1093/eurjhf/hfr090. Epub 2011 Jul 28. PMID 21803755
- [Background] Parati G, Malfatto G, Boarin S, Branzi G, Caldara G, Giglio A, Bilo G, Ongaro G, Alter A, Gavish B, Mancia G. Device-guided paced breathing in the home setting: effects on exercise capacity, pulmonary and ventricular function in patients with chronic heart failure: a pilot study. Circ Heart Fail. 2008 Sep;1(3):178-83. doi: 10.1161/CIRCHEARTFAILURE.108.772640. PMID 19808287
- [Background] Reiner R. Integrating a portable biofeedback device into clinical practice for patients with anxiety disorders: results of a pilot study. Appl Psychophysiol Biofeedback. 2008 Mar;33(1):55-61. doi: 10.1007/s10484-007-9046-6. Epub 2008 Feb 20. PMID 18286369
- [Background] Jacobsen PB, Jim HS. Psychosocial interventions for anxiety and depression in adult cancer patients: achievements and challenges. CA Cancer J Clin. 2008 Jul-Aug;58(4):214-30. doi: 10.3322/CA.2008.0003. Epub 2008 Jun 16. PMID 18558664
- [Background] Mehta KM, Yaffe K, Brenes GA, Newman AB, Shorr RI, Simonsick EM, Ayonayon HN, Rubin SM, Covinsky KE. Anxiety symptoms and decline in physical function over 5 years in the health, aging and body composition study. J Am Geriatr Soc. 2007 Feb;55(2):265-70. doi: 10.1111/j.1532-5415.2007.01041.x. PMID 17302665
- [Background] Schneider S, Moyer A, Knapp-Oliver S, Sohl S, Cannella D, Targhetta V. Pre-intervention distress moderates the efficacy of psychosocial treatment for cancer patients: a meta-analysis. J Behav Med. 2010 Feb;33(1):1-14. doi: 10.1007/s10865-009-9227-2. Epub 2009 Sep 27. PMID 19784868
- [Background] Weaver KE, Forsythe LP, Reeve BB, Alfano CM, Rodriguez JL, Sabatino SA, Hawkins NA, Rowland JH. Mental and physical health-related quality of life among U.S. cancer survivors: population estimates from the 2010 National Health Interview Survey. Cancer Epidemiol Biomarkers Prev. 2012 Nov;21(11):2108-17. doi: 10.1158/1055-9965.EPI-12-0740. Epub 2012 Oct 30. PMID 23112268
- [Background] Burris JL, Andrykowski M. Disparities in mental health between rural and nonrural cancer survivors: a preliminary study. Psychooncology. 2010 Jun;19(6):637-45. doi: 10.1002/pon.1600. PMID 19582800
- [Background] Hewitt M, Greenfield S, Stovall E. From cancer patient to cancer survivor: Lost in Transition. 2006. National Academies Press.
- [Background] Stamm BH, Piland NF, Lambert D, Speck NC. A Rural Perspective on Health Care for the Whole Person. Professional Psychology: Research and Practice 2007;38(3):298-304
- [Background] American Psychological Association, Practice Directorate, Office of Rural Health (2002a). Caring for the rural community: 2000-2001 report. Washington, DC: APA Press; 2001.
- [Background] Jerath R, Edry JW, Barnes VA, Jerath V. Physiology of long pranayamic breathing: neural respiratory elements may provide a mechanism that explains how slow deep breathing shifts the autonomic nervous system. Med Hypotheses. 2006;67(3):566-71. doi: 10.1016/j.mehy.2006.02.042. Epub 2006 Apr 18. PMID 16624497
- [Background] Carrieri-Kohlman V, Gormley JM, Douglas MK, Paul SM, Stulbarg MS. Exercise training decreases dyspnea and the distress and anxiety associated with it. Monitoring alone may be as effective as coaching. Chest. 1996 Dec;110(6):1526-35. doi: 10.1378/chest.110.6.1526. PMID 8989072
- [Background] Gallo-Silver L, Pollack B. Behavioral interventions for lung cancer-related breathlessness. Cancer Pract. 2000 Nov-Dec;8(6):268-73. doi: 10.1046/j.1523-5394.2000.86005.x. PMID 11898143
- [Background] Tanaka K, Akechi T, Okuyama T, Nishiwaki Y, Uchitomi Y. Development and validation of the Cancer Dyspnoea Scale: a multidimensional, brief, self-rating scale. Br J Cancer. 2000 Feb;82(4):800-5. doi: 10.1054/bjoc.1999.1002. PMID 10732749
- [Background] Dudgeon DJ, Lertzman M. Dyspnea in the advanced cancer patient. J Pain Symptom Manage. 1998 Oct;16(4):212-9. doi: 10.1016/s0885-3924(98)00065-7. PMID 9803048
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Luckett T, Butow PN, King MT, Oguchi M, Heading G, Hackl NA, Rankin N, Price MA. A review and recommendations for optimal outcome measures of anxiety, depression and general distress in studies evaluating psychosocial interventions for English-speaking adults with heterogeneous cancer diagnoses. Support Care Cancer. 2010 Oct;18(10):1241-62. doi: 10.1007/s00520-010-0932-8. Epub 2010 Jul 2. PMID 20596731
- [Background] Dyspnea. Mechanisms, assessment, and management: a consensus statement. American Thoracic Society. Am J Respir Crit Care Med. 1999 Jan;159(1):321-40. doi: 10.1164/ajrccm.159.1.ats898. No abstract available. PMID 9872857
- [Background] Polanski J, Chabowski M, Chudiak A, Uchmanowicz B, Janczak D, Rosinczuk J, Mazur G. Intensity of Anxiety and Depression in Patients with Lung Cancer in Relation to Quality of Life. Adv Exp Med Biol. 2018;1023:29-36. doi: 10.1007/5584_2017_50. PMID 28573442
- [Background] Krebber AM, Jansen F, Witte BI, Cuijpers P, de Bree R, Becker-Commissaris A, Smit EF, van Straten A, Eeckhout AM, Beekman AT, Leemans CR, Verdonck-de Leeuw IM. Stepped care targeting psychological distress in head and neck cancer and lung cancer patients: a randomized, controlled trial. Ann Oncol. 2016 Sep;27(9):1754-60. doi: 10.1093/annonc/mdw230. Epub 2016 Jun 10. PMID 27287209
- [Background] Quist M, Langer SW, Rorth M, Christensen KB, Adamsen L. "EXHALE": exercise as a strategy for rehabilitation in advanced stage lung cancer patients: a randomized clinical trial comparing the effects of 12 weeks supervised exercise intervention versus usual care for advanced stage lung cancer patients. BMC Cancer. 2013 Oct 14;13:477. doi: 10.1186/1471-2407-13-477. PMID 24124893
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510
- [Background] Gift AG. Validation of a vertical visual analogue scale as a measure of clinical dyspnea. Rehabil Nurs. 1989 Nov-Dec;14(6):323-5. doi: 10.1002/j.2048-7940.1989.tb01129.x. PMID 2813949
- [Background] Mancini I, Body JJ. Assessment of dyspnea in advanced cancer patients. Support Care Cancer. 1999 Jul;7(4):229-32. doi: 10.1007/s005200050254. PMID 10423048
- [Background] Kalauokalani D, Cherkin DC, Sherman KJ, Koepsell TD, Deyo RA. Lessons from a trial of acupuncture and massage for low back pain: patient expectations and treatment effects. Spine (Phila Pa 1976). 2001 Jul 1;26(13):1418-24. doi: 10.1097/00007632-200107010-00005. PMID 11458142
- [Background] Linde K, Witt CM, Streng A, Weidenhammer W, Wagenpfeil S, Brinkhaus B, Willich SN, Melchart D. The impact of patient expectations on outcomes in four randomized controlled trials of acupuncture in patients with chronic pain. Pain. 2007 Apr;128(3):264-271. doi: 10.1016/j.pain.2006.12.006. Epub 2007 Jan 25. PMID 17257756
- [Background] Cancer of the Lung and Bronchus - SEER Stat Fact Sheets [Internet]. [cited 2012 Jul 17]. Available from: http://seer.cancer.gov/statfacts/html/lungb.html
- [Background] Simon R, Wittes RE, Ellenberg SS. Randomized phase II clinical trials. Cancer Treat Rep. 1985 Dec;69(12):1375-81. PMID 4075313
- [Background] Wilson EB. Probable inference, the law of succession, and statistical inference. JASA1927;22: 209-212.
- [Background] Garcia SF, George J, Rosenbloom SK, Cella D. Adapting chronic illness health related quality of life item banks for cancer populations. In Poster presented at the International Society for Quality of LifeResearch on Patient-Reported Outcomes in Clinical Practice, Budapest, Hungary. In 2007.
- [Background] Molassiotis A, Ellis J, Wagland R, Williams ML, Bailey CD, Booton R, Blackhall F, Yorke J, Smith JA. The Manchester cough in lung cancer scale: the development and preliminary validation of a new assessment tool. J Pain Symptom Manage. 2013 Feb;45(2):179-90. doi: 10.1016/j.jpainsymman.2012.01.015. Epub 2012 Aug 25. PMID 22926094
- [Background] Uddin M, Aiello AE, Wildman DE, Koenen KC, Pawelec G, de Los Santos R, Goldmann E, Galea S. Epigenetic and immune function profiles associated with posttraumatic stress disorder. Proc Natl Acad Sci U S A. 2010 May 18;107(20):9470-5. doi: 10.1073/pnas.0910794107. Epub 2010 May 3. PMID 20439746
- [Background] Uddin M, Koenen KC, Aiello AE, Wildman DE, de los Santos R, Galea S. Epigenetic and inflammatory marker profiles associated with depression in a community-based epidemiologic sample. Psychol Med. 2011 May;41(5):997-1007. doi: 10.1017/S0033291710001674. Epub 2010 Sep 14. PMID 20836906
- [Background] El-Sayed AM, Haloossim MR, Galea S, Koenen KC. Epigenetic modifications associated with suicide and common mood and anxiety disorders: a systematic review of the literature. Biol Mood Anxiety Disord. 2012 Jun 14;2:10. doi: 10.1186/2045-5380-2-10. PMID 22738307
- [Background] Weaver IC, Cervoni N, Champagne FA, D'Alessio AC, Sharma S, Seckl JR, Dymov S, Szyf M, Meaney MJ. Epigenetic programming by maternal behavior. Nat Neurosci. 2004 Aug;7(8):847-54. doi: 10.1038/nn1276. Epub 2004 Jun 27. PMID 15220929
- [Background] Aldwin, C M, The physiology of stress, in Stress, Coping, and Development Guilford Press: New York, NY. 2007; 39-54.
- [Background] Murphy SE, Braithwaite EC, Hubbard I, Williams KV, Tindall E, Holmes EA, Ramchandani PG. Salivary cortisol response to infant distress in pregnant women with depressive symptoms. Arch Womens Ment Health. 2015 Apr;18(2):247-253. doi: 10.1007/s00737-014-0473-0. Epub 2014 Oct 29. PMID 25352317
- [Background] Schrepf A, Clevenger L, Christensen D, DeGeest K, Bender D, Ahmed A, Goodheart MJ, Dahmoush L, Penedo F, Lucci JA 3rd, Ganjei-Azar P, Mendez L, Markon K, Lubaroff DM, Thaker PH, Slavich GM, Sood AK, Lutgendorf SK. Cortisol and inflammatory processes in ovarian cancer patients following primary treatment: relationships with depression, fatigue, and disability. Brain Behav Immun. 2013 Mar;30 Suppl(0):S126-34. doi: 10.1016/j.bbi.2012.07.022. Epub 2012 Aug 5. PMID 22884960
- [Background] Stoppelbein L, Greening L. A longitudinal study of the role of cortisol in posttraumatic stress disorder symptom clusters. Anxiety Stress Coping. 2015;28(1):17-30. doi: 10.1080/10615806.2014.923844. Epub 2014 Jun 17. PMID 24824647
- [Background] Vadiraja HS, Raghavendra RM, Nagarathna R, Nagendra HR, Rekha M, Vanitha N, Gopinath KS, Srinath BS, Vishweshwara MS, Madhavi YS, Ajaikumar BS, Ramesh BS, Nalini R, Kumar V. Effects of a yoga program on cortisol rhythm and mood states in early breast cancer patients undergoing adjuvant radiotherapy: a randomized controlled trial. Integr Cancer Ther. 2009 Mar;8(1):37-46. doi: 10.1177/1534735409331456. Epub 2009 Feb 3. PMID 19190034
- [Background] Cruess DG, Antoni MH, McGregor BA, Kilbourn KM, Boyers AE, Alferi SM, Carver CS, Kumar M. Cognitive-behavioral stress management reduces serum cortisol by enhancing benefit finding among women being treated for early stage breast cancer. Psychosom Med. 2000 May-Jun;62(3):304-8. doi: 10.1097/00006842-200005000-00002. PMID 10845343
- [Background] Nickel C, Tanca S, Kolowos S, Pedrosa-Gil F, Bachler E, Loew TH, Gross M, Rother WK, Nickel MK. Men with chronic occupational stress benefit from behavioural/psycho-educational group training: a randomized, prospective, controlled trial. Psychol Med. 2007 Aug;37(8):1141-9. doi: 10.1017/S0033291706009445. Epub 2006 Dec 6. PMID 17147835
- [Background] Boyes A, D'Este C, Carey M, Lecathelinais C, Girgis A. How does the Distress Thermometer compare to the Hospital Anxiety and Depression Scale for detecting possible cases of psychological morbidity among cancer survivors? Support Care Cancer. 2013 Jan;21(1):119-27. doi: 10.1007/s00520-012-1499-3. Epub 2012 May 24. PMID 22618735
- [Background] Donovan KA, Grassi L, McGinty HL, Jacobsen PB. Validation of the distress thermometer worldwide: state of the science. Psychooncology. 2014 Mar;23(3):241-50. doi: 10.1002/pon.3430. Epub 2013 Nov 11. PMID 25160838
- [Background] Ma X, Zhang J, Zhong W, Shu C, Wang F, Wen J, Zhou M, Sang Y, Jiang Y, Liu L. The diagnostic role of a short screening tool--the distress thermometer: a meta-analysis. Support Care Cancer. 2014 Jul;22(7):1741-55. doi: 10.1007/s00520-014-2143-1. Epub 2014 Feb 8. PMID 24510195
- [Background] Custers JA, van den Berg SW, van Laarhoven HW, Bleiker EM, Gielissen MF, Prins JB. The Cancer Worry Scale: detecting fear of recurrence in breast cancer survivors. Cancer Nurs. 2014 Jan-Feb;37(1):E44-50. doi: 10.1097/NCC.0b013e3182813a17. PMID 23448956
- [Derived] Danhauer SC, Dressler EV, Brown WM, Nightingale CL, Brenes GA, Petty WJ, Curtis A, Murkutla S, Huang J, Wagi CR, Lesser GJ, Weaver KE. Reducing Anxiety and Dyspnea via Device-Guided Breathing (RELAX): A Multi-Site Feasibility Study in Post-Treatment Lung Cancer Survivors at Community Cancer Clinics (WF-01213). Integr Cancer Ther. 2023 Jan-Dec;22:15347354231164406. doi: 10.1177/15347354231164406. PMID 37029555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Implementation was facilitated through the Wake Forest National Cancer Institute Community Oncology Research Program (NCORP), developed to increase community participation in cancer trials. Forty-six participants were accrued between July 30 2015 and June 11 2019 (0.99 participants/month).
Pre-assignment Details: In this feasibility study, participants were stratified by baseline self-reported dyspnea score and randomized to a 12-week high-dose or low-dose device-guided breathing intervention versus a usual breathing control group with equal probability, using variable length permuted block randomization. All participants enrolled were randomized and included in analyses.
Groups:
- Group A - Device Guided Breathing Low Dose. 15 Minutes Once a Day, 5 Days a Week for 12 Weeks.: Group A - Device Guided Breathing Low Dose
  Group A - Device guided breathing low dose: Group A: 15 minutes once a day, 5 days a week for 12 weeks.
- Group B - Device Guided Breathing High Dose. 15 Minutes Twice a Day, 5 Days a Week for 12 Weeks.: Group B - Device guided breathing high dose
  Group B - Device guided breathing high dose: Group B - 15 minutes twice a day, 5 days a week for 12 weeks.
- Group C - Usual Breathing Control Group. 15 Minutes Per Day, 5 Days a Week for 12 Weeks.: Group C - Usual Breathing Control Group
  Group C - Usual Breathing Control Group: Group C - 15 minutes per day, 5 days a week for 12 weeks.
Period: Overall Study
Arm/Group | Group A - Device Guided Breathing Low Dose. 15 Minutes Once a Day, 5 Days a Week for 12 Weeks. | Group B - Device Guided Breathing High Dose. 15 Minutes Twice a Day, 5 Days a Week for 12 Weeks. | Group C - Usual Breathing Control Group. 15 Minutes Per Day, 5 Days a Week for 12 Weeks.
Started | 14 | 14 | 18
Week 6 | 11 | 9 | 14
Completed | 10 | 8 | 14
Not Completed | 4 | 6 | 4
Not completed — Withdrawal by Subject | 4 | 6 | 3
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 14 | 14 | 18 | 46
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 76] | 64 [41 to 77] | 66 [43 to 74] | 65 [41 to 77]
Age, Customized [Count of Participants; unit: Participants]
  Age: >=50 years | 13 | 11 | 17 | 41
  Age: <50 | 1 | 3 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 13 | 35
  Male | 4 | 2 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 18 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 6
  White | 10 | 12 | 14 | 36
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 18 | 46
Cancer Dyspnea Scale [Count of Participants; unit: Participants] — 12-item self-report measure of multidimensional (sense of effort, sense of anxiety, discomfort) nature of dyspnea. Reliable and valid in lung cancer patients. Scores range from 0-44 and clinical dyspnea is considered total scores greater than or equal to 8. Higher scores reflect more dyspnea. Selected as an optimal measure of dyspnea since it assesses multiple symptom components and is validated for use in cancer survivors.
  Participants
    <8 | 6 | 6 | 9 | 21
    >=8 | 8 | 8 | 9 | 25
Marital Status [Count of Participants; unit: Participants]
  Single | 0 | 0 | 0 | 0
  Married | 8 | 8 | 13 | 29
  Separated/Divorced/Widowed | 6 | 6 | 2 | 14
  Unknown | 0 | 0 | 3 | 3
Income [Count of Participants; unit: Participants]
  Under $20,000 | 4 | 2 | 6 | 12
  $20,000 - $49,999 | 5 | 5 | 8 | 18
  $50,000 or more | 2 | 5 | 2 | 9
  Unknown | 3 | 2 | 2 | 7
Education [Count of Participants; unit: Participants]
  High School or Less | 2 | 0 | 1 | 3
  College graduate or some college | 10 | 9 | 13 | 32
  Post College Graduate Education | 2 | 5 | 4 | 11
Stage of Disease [Count of Participants; unit: Participants] — Clinical staging of the disease based on the American Joint Committee on Cancer (AJCC) system. Ranges from 0 to IV with higher numbers reflecting more severe disease. In non-small cell lung cancer stage 0 is where the tumor is found only in the top layers of cells lining the air passages, but it has not invaded deeper into other lung tissues to stage IV where it has spread to the other lung or other areas of the body.
  Participants
    I | 2 | 6 | 7 | 15
    II | 2 | 1 | 2 | 5
    III | 3 | 4 | 1 | 8
    IV | 7 | 3 | 8 | 18
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Standardizes how the disease impacts a patient's daily living abilities. Scale ranges from 0 to 5. Higher scores are worse. 0-Fully active, able to carry on all pre-disease performance without restriction; 1-Restricted in physically strenuous activity but ambulatory and able to carry out light/sedentary work; 2-Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about >50% waking hours; 3-Capable of only limited selfcare; confined to bed or chair >50% waking hours; 4-Completely disabled; cannot carry on any selfcare; totally confined to bed/chair; 5-Dead
  Participants
    0 | 6 | 6 | 6 | 18
    1 | 8 | 7 | 8 | 23
    2 | 0 | 1 | 4 | 5
Current Smoker [Count of Participants; unit: Participants]
  Yes | 2 | 4 | 4 | 10
  No | 12 | 10 | 14 | 36

OUTCOME MEASURES:

1. Primary Outcome: Retention - Number of Participants Who Complete the Final Assessment
Description: Retention will be calculated as the number of participants who complete the final assessment divided by number randomized.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 14 | 18
Participants | 10 | 8 | 14

2. Primary Outcome: Adherence- Amount of Time the Device is Used
Description: Adherence will be calculated as the actual amount of time the device is used divided by the prescribed time. Successful adherence will be defined as use of the device ≥80% of the time assigned.
Time Frame: 12 weeks
Population: Adherence data used visits up to withdrawal or study completion. Includes 5 participants missing all breathing visits. Excludes 2 participants that withdrew at baseline and have no available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 13 | 13 | 18
Participants
  Overall | 13 | 8 | 12
  Weeks 1-6 | 13 | 9 | 14
  Weeks 7-12: number analyzed (Participants) | 11 | 10 | 16
  Weeks 7-12 | 10 | 6 | 11

3. Primary Outcome: Accrual Rate- Number of Patients Accrued to the Study
Description: The accrual rate will be calculated as the number of patients accrued to the study divided by the number of months of accrual.
Time Frame: Time from study opening to study close ~46.42 months
Population: Participants were accrued between July 30 2015 and June 11 2019 for a total of 46.42 months.
Measure: Number; unit: participants per month
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 14 | 18
participants per month | 0.30 | 0.30 | 0.39

4. Secondary Outcome: Change From Baseline for Anxiety as Measured by Hospital Anxiety and Depression Scale (HADS)
Description: To obtain preliminary data on the variability and efficacy of two doses of a device-guided breathing intervention versus a usual breathing control group for reducing anxiety. This is a 14-item self-report measure of cognitive and behavioral symptoms of anxiety and depression; clinically significant symptoms are indicated by a score of greater than or equal to 8 with a range from 0 to 42. Higher scores indicate more anxiety.
Time Frame: 12 weeks
Population: All data was utilized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 14 | 18
score on a scale
  Change from baseline to 6 weeks | -1.22 [-2.90 to 0.45] | -2.38 [-4.34 to -0.43] | -1.75 [-3.21 to -0.29]
  Change from baseline to 12 weeks | -2.27 [-3.55 to -0.99] | -2.10 [-3.74 to -0.45] | -1.89 [-3.01 to -0.77]

5. Other Pre Specified Outcome: Salivary Cortisol Levels
Description: Cortisol levels will be assessed upon awakening, 30 minutes post-awakening, and at bedtime for three consecutive days at baseline and three consecutive days.
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: DNA Methylation Levels
Description: DNA methylation levels will be measured To determine if changes in anxiety are associated with methylation
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Gene Expression Levels
Description: The DNA methylation and gene expression patterns between the different groups.
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Event/Serious Adverse Event reporting begins after the informed consent is signed and is followed for 30 days post study completion, an average of 16 weeks
Description: Only report unexpected serious adverse events, Grades 4 and 5, which are related to the use of the breathing device used in this study. Serious Adverse Events occurring within 30 days of study completion must be reported via FDA Form 3500 (MedWatch).
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 1/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/18

LIMITATIONS AND CAVEATS:
Trial terminated early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT02063828/Prot_SAP_001.pdf
  • Informed Consent Form (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT02063828/ICF_002.pdf